CLINICAL TRIAL: NCT07296042
Title: Targeted And Perilesional Or Systematic Biopsy In Prostate Cancer
Acronym: TARGET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COS-RGDS-2025-06-003-TARGET; 2025-A02500-49 (Other: IDRCB)
Record Dates: First submitted 2025-11-14; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: MRI; biopsy; prostate cancer detection; clinically significant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Each patient will be its own control as each patient will receive targeted, regional and systematic biopsies of the prostate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New prostate biopsy scheme (Other): Control and experimental performed in the same arm
  Interventions: Procedure: Prostate biopsy

INTERVENTIONS:
Procedure: Prostate biopsy — The intervention for this study will be a modification of the standard prostate biopsy scheme. Instead of a targeted + systematic biopsy (3 targeted and 12 systematic biopsies (6 in each lobe)), the following 15 biopsies will be performed:
  * 3 targeted biopsies
  * 4 regional biopsies
  * 8 systematic biopsies (2 posterior right, 2 lateral right, 2 posterior left, 2 lateral left)

SUMMARY:
Magnetic Resonance Imaging (MRI) improves the detection of clinically significant prostate cancer (PCa) by guiding biopsies of MRI-visible lesions (targeted biopsies) in patients suspected with having PCa. This strategy increases the detection of clinically significant PCa, however, while also increasing the detection of insignificant prostate cancer, often synonymous of "overdiagnosis".

It is well known that insignificant PCa has a very low risk of local and distant progression, and active surveillance with a deferred curative treatment protocol based on clear indicators of disease progression is now recommended for all insignificant PCa. However, higher detection of insignificant PCa can lead to patient anxiety about inclusion in an active surveillance protocol, potential further damage from repeated surveillance biopsies and higher healthcare costs.

Thus, there is a need for a new biopsy scheme that maintains clinically significant PCa's detection while reducing the diagnosis of insignificant PCa. In recent years, an alternative approach has been to add additional cores close to the target lesion, this is defined as regional biopsies. The hypothesis is that most clinically significant PCa missed in the target are found close to the target. Whereas most cancers found on systematic biopsies outside the MRI target probably correspond to insignificant PCa. This strategy aims to maintain the detection of clinically significant PCa, while reducing the detection of insignificant PCa.

This proposed multicenter diagnostic study aims to demonstrate the effectiveness of the experimental biopsy scheme (targeted + regional) in detecting clinically significant PCa, compared with a conventional scheme (targeted + systematic). We also aim to compare the detection of insignificant PCa by both schemes.

DETAILED DESCRIPTION:
In prostate cancer (PCa), the descriptor 'clinically significant' is widely used to differentiate PCa that may cause morbidity or death in a specific patient from types of PCa that rarely do. The definition of significant vs. insignificant is a balance between tumor and patient factors. In current guidelines and literature, it is widely accepted that insignificant PCa corresponds to almost all men with an International Society of Urological Pathology (ISUP) grade group 1, while clinically significant PCa is defined as any ISUP grade group ≥2.

This distinction is particularly important as insignificant PCa is more common than significant PCa. The detection of insignificant PCa has increased since the introduction of the prostate-specific antigen (PSA) test in the 1990s, and poses several problems of over-diagnosis and over-treatment, considered to be major drawbacks of population-wide screening and individual early detection. It is well known that insignificant PCa has very low risk of local and distant progression, and an active surveillance associated with a deferred curative treatment protocol based on clear indicators of disease progression, is now recommended for all insignificant PCa. However, higher detection of insignificant PCa can lead to patient anxiety about inclusion in an active surveillance protocol, potential further damage from repeated surveillance biopsies and higher healthcare costs. Therefore, our objective during PCa screening is to maintain the detection of clinically significant PCa while decreasing the diagnosis of insignificant PCa.

Magnetic Resonance Imaging (MRI) is currently indicated prior to prostate biopsy and is used to identify and locate suspicious lesions for clinically significant PCa. Indeed, correlation with radical prostatectomy specimens shows that MRI has good sensitivity for the detection and localization of ISUP grade group ≥ 2 PCa. Several recent large-scale randomized controlled trials have shown that pre-biopsy MRI and MRI-targeted biopsy are the best modality for increasing the detection of clinically significant PCa, while reducing the detection of clinically insignificant PCa, in comparison with a systematic biopsy scheme.

Radiologists use multi-level scoring systems according to the Likert scale principle; where the presence of clinically significant prostate cancer in a lesion can be subjectively categorized as highly unlikely to highly likely, with a varying number of subdivisions. The 1 to 5 scale according to the Prostate Imaging - Reporting and Data System (PI-RADS) version 2.1 provides guidance for radiologists with more objective criteria and is currently most often used.

The PI-RADS score is used in clinical practice as a triage test to indicate the need for prostate biopsy. Patients with a PI-RADS score of 1 or 2 have a very low risk of having clinically significant PCa (<5%), and prostate biopsy is generally not performed in these cases to avoid diagnosing insignificant PCa (20%). The same principle applies to patients with a PI-RADS 3 lesion. In a multicenter cohort of 1476 men with PI-RADS 3 lesions, the prevalence of ISUP grade group ≥ 2 was 18.5%. Applying a PSA density cut-off of 0.15 ng/mL/cc, 817 biopsy procedures (58.4%) would have been avoided at the cost of missing ISUP grade group ≥ 2 PCa in only 91 men (6.5%) and ISUP grade group 1 PCa would not have been detected in 115 men (8.2%). Consequently, current guidelines recommend avoiding biopsy in patients with a PI-RADS 3 lesion and low PSA density. In patients with a PI-RADS 4 or 5 lesion, prostate biopsy is strongly indicated, as the prevalence of clinically significant PCa ranges from 31% to 77%.

Despite recent advances in MRI, the current recommended prostate biopsy scheme, i.e., targeted + systematic biopsy, leads to a 5.8% increase in the detection of clinically significant PCa, at the cost of a 15% increase in insignificant PCa. There is therefore still over-diagnosis of insignificant PCa. This over-diagnosis of insignificant PCa is largely attributed to systematic biopsies, where the operator takes a sample from the prostatic lobe that is not suspicious on MRI. Today, the need to perform systematic biopsies in association with targeted biopsies is strongly questioned. However, targeted only biopsies significantly underperform targeted + systematic biopsies in detecting significant PCa.

In light of this, the PI-RADS Committee recently introduced the concept of "penumbra" and recommended the addition of regional sampling to the targeted biopsies. In fact, most clinically significant PCa (>90%) missed by targeted biopsies are found within a 10-mm radius of the MRI-visible lesion. Including additional regional biopsies, rather than standard sextant-based systematic biopsies may decrease the total number of cores taken (by avoiding systematic biopsies in MRI-negative lobes) and improve the detection of clinically significant PCa (by compensating for guiding imprecision). In addition, the MRI-targeted and regional biopsy approach could avoid detecting 12-17% of the insignificant PCa detected by the classical targeted + systematic approach. These findings are corroborated by a very recent systematic review and meta-analysis comparing the two approaches: systematic + targeted biopsy vs. regional + targeted biopsy. This meta-analysis revealed a non-statistically significant increase in the detection of clinically significant PCa in the regional + targeted biopsy group (46.1% vs. 44.2%; odds ratio [OR] 1.07, 95% confidence interval [CI] 0.99-1.16, p=0.07) compared with the standard biopsy scheme. Furthermore, compared with a regional biopsy scheme, systematic biopsies led to an increase in the detection of insignificant PCa (OR 1.16, 95% CI 1.04-1.30, p=0.008).

While this new biopsy scheme (i.e. targeted + regional) looks promising, there are several limitations that need to be recognized. First, most published data are based on retrospective studies, and high-quality data from prospective studies are lacking. Second, all studies are based on a targeted + systematic biopsy scheme, and regional biopsies were retrospectively identified as systematic cores taken close to the MRI index lesion. Third, there is no standardization of regional biopsy sampling, with some authors taking cores within 10 mm, 15 mm, 20 mm of the lesion visible on MRI, or even sampling the entire lobe ipsilateral to the lesion without any consensus. All these limitations, and mainly the lack of prospective validation, led us not to recommend this approach in our latest French guidelines.

Brisbane et al. found that more than 90% of non-targeted biopsies containing clinically significant PCa cores were found within a 10-mm radius of the MRI-visible lesion. While a few cores containing clinically significant cancer were located outside the 10 mm radius, yield decreased with increasing distance from the zone of interest. Therefore, regional biopsies are usually performed within a 10-mm radius of the MRI-visible lesion. Optimal placement and numbers of targeted and regional biopsies are yet to be determined. Previous studies seem to suggest that a minimum of 3-4 biopsy cores per zone is necessary to overcome sampling errors and maintain optimal detection of clinically significant PCa. Based on these results, the ideal scheme for regional biopsy appears to be 3-4 cores within a 10 mm radius of the index lesion. In the TARGET trial, before the first inclusion, an investigators' meeting will be organized to ensure homogeneity of the biopsy technique applied.

ELIGIBILITY:
Inclusion Criteria:

* Adult men (≥ 18 years old)
* Clinical suspicion of PCa (based on digital rectal examination, family history, PSA and PSA density values) and prescribed prostate biopsy
* Detection by multi-parametric MRI of the prostate of a PI-RADS 4 or 5 index lesion, or a PI-RADS 3 index lesion with a PSA density ≥ 0.15 ng/ml/cc
* Patient eligible for prostate biopsy under local or general anesthesia
* PSA ≤ 20 ng/mL
* Patient who agreed to participate in the study and signed the consent form

Exclusion Criteria:

* History of prostate cancer
* History of negative prostate biopsy
* MRI negative (PI-RADS 1 or 2) or equivocal (PI-RADS 3) with PSA density < 0.15 ng/ml/cc
* Patient unable to understand the terms of the study or unable to give informed consent (neurological or psychiatric disorders, non-French speaker, etc.)
* Patient under full or partial legal guardianship.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the targeted + regional biopsy scheme for the detection of clinically significant prostate cancer | On the day of the biopsy (up to day 90)
  The primary endpoint is the sensitivity and specificity of the targeted + regional biopsy scheme for the detection of clinically significant PCa (ISUP grade group ≥ 2) compared to the sensitivity and specificity of the targeted + systematic biopsy scheme (standard of care).
  A biopsy will be considered negative if there is no cancer or only insignificant PCa (ISUP grade 1 group) detected. A biopsy will be considered positive if there is clinically significant PCa (ISUP grade ≥ 2 group) detected.

SECONDARY OUTCOMES:
Detection of not significant prostate cancer | On the day of the biopsy (up to day 90)
  Difference in the detection rate of insignificant PCa (ISUP grade group 1) depending on the biopsy scheme (experimental vs standard)
Detection of agressive prostate cancer | On the day of the biopsy (up to day 90)
  Difference in the detection rate of aggressive PCa (ISUP grade group ≥ 3) depending on the biopsy scheme (experimental vs standard)
Creation of a nomogram for the detection of clinically significant prostate cancer | On the day of the biopsy (up to day 90)
  The endpoint of the nomogram is the detection of clinically significant PCa using a targeted + regional biopsy scheme

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Nord, Assistance Publique des Hôpitaux de Marseille, Marseille
  - CHI Mont de Marsan - Site de Layné, Mont-de-Marsan
  - Hôpital privé des Peupliers - Ramsay Santé, Paris
  - Clinique La Croix du Sud - RAMSAY Santé, Quint-Fonsegrives

IPD SHARING:
Plan to Share IPD: Undecided